CLINICAL TRIAL: NCT04911036
Title: Study of the Effect of the Time of Diagnosis (Antenatal vs. Postnatal) on the Post-traumatic Reactions of Parents of Children Undergoing Oesophageal Atresia Surgery "
Acronym: DANAO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_26; 2020-A00255-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atresia, Esophageal
Keywords: Esophageal atresia; post-traumatic reactions; early accompaniment; Perinatal Posttraumatic Stress Disorder Questionnaire; cross-sectional study in psychology
MeSH Terms: conditions — Esophageal Atresia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers and/or fathers with an antenatal diagnosis
  Interventions: Other: Questionnaires
- Mothers and/or fathers with a postnatal diagnosis
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Perinatal PTSD Questionnaire State Trait Anxiety Inventory-forme Y-B Early Support Questionnaire Socio-demographic questionnaire

SUMMARY:
This is an observational, national multicentre (34 centres involved), cross-sectional study in psychology whose objective is to describe and compare the levels of post-traumatic reactions of mothers to the announcement of their child's EA diagnosis.

An ancillary study will be carried out among the fathers present who agree to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Be the mother and/or a father of a living child aged 12 to 24 months who has undergone neonatal surgery following the diagnosis of type 1 or type 3 EA;
* Not to have objected to participating in the study (information and non-objection form signed by the investigator);
* To be socially insured.

Exclusion Criteria:

* Woman or man whose child with AO has a chromosomal abnormality;
* Woman or man whose child with AO has a polymalformative syndrome;
* Female or male minor ;
* Pregnant woman;
* Woman or man who does not speak French;
* Woman or man unable to consent, or benefiting from a legal protection regime (guardianship or curatorship);
* Woman or man deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Be a mother and/or a father of a living child aged between 12 and 24 months who has undergone neonatal surgery following a diagnosis of type 1 or type 3 EA
Study Population: Be a mother and/or a father of a living child aged between 12 and 24 months who has undergone neonatal surgery following a diagnosis of type 1 or type 3 EA
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Perinatal Posttraumatic Stress Disorder Questionnaire (score PPQ) | at 2 months
  The score PPQ derived from this instrument corresponds to the number of items (there are 14) to which the parent responded positively (theoretical spread: 0-14 points)

SECONDARY OUTCOMES:
Percentage of mothers with Score PPQ >5 | at 2 months
Questionnaire on early support | at 2 months
  This is a questionnaire co-constructed with the Association Française de l'Atresie de l'œsophage (AFAO) to collect information on the perception of support available or received upon suspicion of an abnormality in the child. It consists of 15 questions. The first eight explore satisfaction with various aspects of early support (information, support, professionals met...). The next seven address parental perceptions regarding information and support. Most of the questions are to be answered on a 5-point Likert scale (e.g., from "Not at all satisfied" to "Very satisfied" or "Never" to "Almost always"), the other questions are closed-ended. Time to complete the test: 5 to 10 minutes.
Correlation between STAI-Trait, Questionnaire on early support and Score PPQ evaluated to mothers | at 2 months
  State-Trait Anxiety Inventory (STAI-TRAIT) SCORE: 20 items in the form of a 4-response Likert scale (from 1 : low anxiety to 4 : highest anxiety). The score goes from 20 to 80 depending of the degree of anxiety.
Correlation between STAI-Trait, Questionnaire on early support and Score PPQ evaluated to fathers | at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Debarge, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France